CLINICAL TRIAL: NCT07297121
Title: Validation of the Montreal Cognitive Assessment (MoCA) Version 8.x and MoCA-MIS in Greece.
Status: Not yet recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: MoCA Clinic and Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 207/2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: MCI; Dementia; Mild Cognitive Impairment (MCI)
Keywords: MCI; MoCA; MoCA-MIS; Validation; Mild Cognitive Impairment; screening; dementia; memory testing
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group
- Group were patients have a MCI diagnosis
- Demented patients

SUMMARY:
Objective: The purpose of this study is to assess the psychometric qualities of the Montreal Cognitive Assessment (MoCA) version 8.x in Greek, including the MoCA-MIS. We intend to examine the tool's reliability (internal consistency, test-retest reliability) and validity (construct validity, concurrent validity, and known-group validity).

Aim: The findings will support the tool's application for early cognitive impairment identification in clinical and research settings.

DETAILED DESCRIPTION:
MoCA is an increasingly common instrument used for cognitive assessment globally. Version 8.x has been translated into Greek, however a validation is of great importance. The participants of this study will be recruited from the outpatient clinic of the 3rd Department of Psychiatry School of Medicine, General University Hospital of Thessaloniki "AHEPA".

The Greek version of MoCA 8.x will be used to evaluate the participants with an analogous cognitive test, such as Addenbrooke's Cognitive Examination (ACE-III) and the M-ACE.

Within 4 weeks, the MoCA will be administered again to a subgroup again in order to evaluate the tool's test-retest reliability. In addition to internal consistency, construct validity (as measured by factor analysis), concurrent validity (correlation with existing tools), and known-group validity (comparing scores between cognitively healthy individuals and those with MCI or dementia), known-group validity will also be evaluated.

Study Type and Time Frames:

Observational Model: Cohort Cross-sectional with a short-timed phase (test-retest). The study is estimated to be completed withing a year's period.

Measure Time Frame Description Internal Consistency Baseline Assessment of internal reliability Test-retest Reliability 4 weeks post-baseline Stability of the test over time Construct Validity Baseline Factor analysis to explore the underlying structure Concurrent Validity Baseline Correlation with established cognitive tools Known-groups Validity Baseline Score comparison across diagnostic groups

Eligibility Criteria:

* Participants between the ages of 55-85
* Fluent in Greek to avoid misunderstandings during the assessment
* Participants must be able to provide informed consent

Exclusion Criteria:

* History of severe psychiatric or neurological disorders apart from MCI/dementia
* Patients having acute medical illnesses
* Patients having severe hearing and/or visual impairments

Study's Population Size:

* 50-100 Cognitively Healthy Adults
* 50-75 MCI Patients
* 50-75 Demented Patients

Location:

Outpatient clinic of the 3rd Department of Psychiatry, School of Medicine, General University Hospital of Thessaloniki "AHEPA", Aristotle University of Thessaloniki, Greece.

Kiriakidi 1, Thessaloniki 546 36 Contact: +302313303110

Principal Investigator:

Dr. Nikitas Arnaoutoglou, MD, PhD Affiliation: Assistant Professor of Psychiatry, 3rd Department of Psychiatry, School of Medicine, General University Hospital of Thessaloniki "AHEPA", Aristotle University of Thessaloniki.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 55-85
* Fluent in Greek to avoid misunderstandings during the assessment
* Participants must be able to provide informed consent

Exclusion Criteria:

* History of severe psychiatric or neurological disorders apart from MCI/dementia
* Patients having acute medical illnesses
* Patients having severe hearing and/or visual impairments

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 50-100 Cognitively Healthy Adults
  * 50-75 MCI Patients
  * 50-75 Demented Patients
  The participants of this study will be recruited from the outpatient clinic of the 3rd Department of Psychiatry School of Medicine, General University Hospital of Thessaloniki "AHEPA".
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The Validation of the Montreal Cognitive Assessment (MoCA) Version 8.x and MoCA-MIS in Greece. | From enrollment to the end of the follow-up period at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic of the 3rd Department of Psychiatry, School of Medicine, General University Hospital of Thessaloniki "AHEPA", Aristotle University of Thessaloniki, Greece., Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh S, Schubert S, Hoon C, Mioshi E, Hodges JR. Validation of the Addenbrooke's Cognitive Examination III in frontotemporal dementia and Alzheimer's disease. Dement Geriatr Cogn Disord. 2013;36(3-4):242-50. doi: 10.1159/000351671. Epub 2013 Aug 15. PMID 23949210
- [Background] Breton A, Casey D, Arnaoutoglou NA. Cognitive tests for the detection of mild cognitive impairment (MCI), the prodromal stage of dementia: Meta-analysis of diagnostic accuracy studies. Int J Geriatr Psychiatry. 2019 Feb;34(2):233-242. doi: 10.1002/gps.5016. Epub 2018 Nov 27. PMID 30370616
- [Background] Julayanont P, Brousseau M, Chertkow H, Phillips N, Nasreddine ZS. Montreal Cognitive Assessment Memory Index Score (MoCA-MIS) as a predictor of conversion from mild cognitive impairment to Alzheimer's disease. J Am Geriatr Soc. 2014 Apr;62(4):679-84. doi: 10.1111/jgs.12742. Epub 2014 Mar 17. PMID 24635004
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019